CLINICAL TRIAL: NCT06407011
Title: Effects of Swedish Massage Prior Circuit Breathing Training on Asthma Control and Respiratory Function in Patients With Asthma
Brief Title: Effects of Swedish Massage Prior Circuit Breathing Training on Asthma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wannaporn Tongtako, Ph.D., Principal investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EX PHYSIO SPSC 10
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Asthma; Status
Keywords: Asthma; Circuit breathing; Swedish massage; Pulmonary function; Asthma control
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Sham Comparator): The CON group did not have any intervention but usual care.
  Interventions: Other: Control
- Swedish massage prior circuit breathing training group (SBT) (Experimental): Participants Swedish massage prior circuit breathing training 3 days/week, 12 weeks. They perform Swedish massage using techniques such as stroking, kneading, and tapping the upper muscle area of the body for 20 minutes per day. Then, they do circuit breathing exercises for about 30 minutes per day, comprising 3 sets of 4 breathing exercises (triflow, power breath, windmill, and balloon blowing), with 1-minute rest between each exercise and 2 minutes between each set.
  Interventions: Other: Swedish massage prior circuit breathing training group (SBT)
- Circuit breathing training group (CBT) (Experimental): Participants perform circuit breathing exercises for about 30 minutes per day, 3 days/week, 12 weeks, comprising 3 sets of 4 breathing exercises (triflow, power breath, windmill, and balloon blowing), with 1-minute rest between each exercise and 2 minutes between each set.
  Interventions: Other: Circuit breathing training group (CBT)

INTERVENTIONS:
Other: Control — The CON group did not have any intervention but usual care.
  Arms: Control
Other: Swedish massage prior circuit breathing training group (SBT) — Participants Swedish massage prior circuit breathing training 3 days/week, 12 weeks. They perform Swedish massage using techniques such as stroking, kneading, and tapping the upper muscle area of the body for 20 minutes per day. Then, they do circuit breathing exercises for about 30 minutes per day, comprising 3 sets of 4 breathing exercises (triflow, power breath, windmill, and balloon blowing), with 1-minute rest between each exercise and 2 minutes between each set.
  Arms: Swedish massage prior circuit breathing training group (SBT)
Other: Circuit breathing training group (CBT) — Participants perform circuit breathing exercises for about 30 minutes per day, 3 days/week, 12 weeks, comprising 3 sets of 4 breathing exercises (triflow, power breath, windmill, and balloon blowing), with 1-minute rest between each exercise and 2 minutes between each set.
  Arms: Circuit breathing training group (CBT)

SUMMARY:
The objective of this study was to determine the effects of Swedish massage prior circuit breathing training on asthma control and respiratory function in patients with asthma.

DETAILED DESCRIPTION:
Thirty patients with asthma aged 20-65 years were randomized into 3 groups: the control group (CON; n=10), the Circuit Breathing Training group (CBT; n=10), and the Swedish Massage prior to Circuit Breathing Training group (SBT; n=10). Participants in the CON group carried out their daily routine without receiving any training program. The CBT group received circuit breathing training sessions lasting thirty minutes each, three times a week for twelve weeks, while the SBT group received a Swedish massage (20 minutes) before circuit breathing exercises (30 minutes) three times a week for twelve weeks. Physiological data, pulmonary function, respiratory muscle strength, cytokine levels, Asthma Control Test scores, Visual Analogue Scale scores, chest expansion, and muscle flexibility variables were analyzed during the pre-test, post-test at 6 weeks, and post-tests at 12 weeks. Two-way repeated measures ANOVA was used to compare the variables between each test and between groups. Statistical significance was defined as p < .05.

ELIGIBILITY:
Inclusion Criteria:

* Being a male or female patient with asthma who is between 20 and 65 years old.
* Being a patient who has been diagnosed by a doctor with asthma for at least 6 months.
* The severity of the disease has been assessed at levels 2 to 4, meaning the volume of air expelled in the first second of breathing quickly and with full force (Forced Expiratory Volume in one second; FEV1) is between 80% and 30% on the date of data collection. This has been certified by a doctor, and the patient is using medication according to the normal treatment plan.
* Must not have other respiratory diseases such as tuberculosis, lung cancer, emphysema, chronic obstructive pulmonary disease (COPD), etc.
* Should not have received exercise training for more than 20 minutes at a time, 3 days/week, or more in the past 6 months before participating in the research.
* Having no communication problems.
* The sample volunteers to participate in the research and agrees to sign the consent form to participate in the research.

Exclusion Criteria:

* Being a patient who has a history of asthma caused by exercise (Exercise-Induced Asthma).
* In case of a force majeure event that makes it impossible to continue participating in the research, such as injury from an accident or illness, etc.
* Participating in less than 80 percent of the training sessions (28 times out of 36 times) for the breathing training group and the group that practiced breathing together with massage.
* Unwillingness to continue participating in the research.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Test : ACT | Change from baseline Asthma Control Test : ACT at 6 and 12 weeks.
  The Asthma Control Test (ACT) consists of 5 questions designed to assess asthma symptoms over the past 4 weeks. A score out of 25 points is given, with a high score indicating good asthma control. A score lower than 20 points indicates that the disease is not well controlled.
The Mini Asthma Quality of Life Questionnaire: Mini AQLQ | Change from baseline The Mini Asthma Quality of Life Questionnaire: Mini AQLQ at 6 and 12 weeks.
  The Mini Asthma Quality of Life Questionnaire (Mini AQLQ) aims to assess changes in life satisfaction related to health status over the past 2 weeks. It consists of a total of 15 questions divided into 4 areas: Signs and symptoms: 5 items, Environmental management: 3 items, Emotion management: 3 items, and Performance of daily activities: 4 items.
Pulmonary function (Forced vital capacity; FVC) | Change from baseline FVC at 6 and 12 weeks.
  The participants were instructed to sit on a chair and wear a nose clip. The researcher provided them with a detailed set of instructions to ensure they performed the maneuver correctly according to guidelines of the American Thoracic Society (ATS). Prior to demonstrating forced inspiration and expiration, the participants were asked to perform three cycles of slow normal breathing as part of the FVC maneuver. FVC will be reported in liter (L).
Pulmonary function (Forced Expiratory Volume in one second; FEV1) | Change from baseline FEV1 at 6 and 12 weeks.
  The participants were instructed to sit on a chair and wear a nose clip. The researcher provided them with a detailed set of instructions to ensure they performed the maneuver correctly according to guidelines of the American Thoracic Society (ATS). Prior to demonstrating forced inspiration and expiration, the participants were asked to perform three cycles of slow normal breathing as part of the FVC maneuver. FEV1 (L) will be reported in liter (L).
Pulmonary function (The ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs; FEV1/FVC) | Change from baseline FEV1/FVC at 6 and 12 weeks.
  The participants were instructed to sit on a chair and wear a nose clip. The researcher provided them with a detailed set of instructions to ensure they performed the maneuver correctly according to guidelines of the American Thoracic Society (ATS). Prior to demonstrating forced inspiration and expiration, the participants were asked to perform three cycles of slow normal breathing as part of the FVC maneuver. FEV1/FVC will be reported in percent (%).
Pulmonary function (Maximal voluntary ventilation; MVV) | Change from baseline MVV at 6 and 12 weeks.
  The participants were instructed to sit on a chair and wear a nose clip. The researcher provided them with a detailed set of instructions to ensure they performed the maneuver correctly according to guidelines of the American Thoracic Society (ATS). During the MVV maneuver, participants were instructed to demonstrate in rapid and forceful inhalation and exhalation for a duration of 10 seconds. MVV will be reported in liter per minute (L/min).
Respiratory muscle strength | Change from baseline Respiratory muscle strength at 6 and 12 weeks.
  Respiratory muscle strength was evaluated by measuring Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) in centimeters of water (cmH2O). The participants were seated and utilized a portable handheld mouth pressure meter (MicroRPM), along with a nose clip. To assess MIP, participants were instructed to exhale until they emptied their lungs at the point of functional residual capacity (FRC). Participants held the device to their mouth and forcefully inhaled for 1-2 seconds. For the measurement of MEP, participants were directed to inhale until their lungs were completely filled with air, starting from the total lung capacity (TLC) point. Participants were asked to maintain the device on their mouth and forcefully exhaled for 1-2 seconds.

SECONDARY OUTCOMES:
Fractional exhaled nitric oxide | Change from baseline Fractional exhaled nitric oxide at 6 and 12 weeks.
  Participants inhaled deeply for two to three seconds before exhaling slowly. Normally, it took 10 seconds to exhale.
Blood chemical data test | Change from baseline concentration of cytokines in serum of interleukin-4 (IL-4), interleukin-5 (IL-5), and interleukin-13 (IL-13) at 6 and 12 weeks.
  Draw 10 milliliters of blood to analyze blood biochemistry, including interleukin-4 (IL-4), interleukin-5 (IL-5), and interleukin-13 (IL-13).
Chest expansion | Change from baseline chest expansion at 6 and 12 weeks.
  The subjects were asked to sit upright with their hands on their hips. They were then asked to exhale fully and inhale fully. The researcher will use a tape measure to measure the expansion of the chest at various levels, including the upper chest at axillary line, midway between the 2nd and 4th ribs, the middle chest at the level of xiphoid process, midway between Ribs 4 - 6, and the lower thorax at the level of the 10th rib.
Trunk flexion | Change from baseline trunk flexion at 6 and 12 weeks.
  Ask the research participant to stand upright. Then, the researcher will take a tape measure and measure the C7 - S1 position and record the measured value. Next, instruct the participants to slowly bend their torso without bending their knees as much as possible, and then read the measurements on the measuring tape and record them.
Trunk extension | Change from baseline trunk extension at 6 and 12 weeks.
  The participants stood up straight, then the researcher took a tape measure and measured the positions C7 - S1, recording the measured values. The subjects were then instructed to slowly stretch their torso as much as possible without stretching their hips or rotating their torso, and then to read the measurement after stretching their back.
Neck flexion | Change from baseline neck flexion at 6 and 12 weeks.
  The participant stood upright, and the researcher placed the goniometer's pivot point over the participant's ear. Then, instruct the participant to slowly bow his or her head with the chin as close to the neck as possible, while placing the goniometer over the tip of the participant's nose. Measure and record the data.
Neck extension | Change from baseline neck extension at 6 and 12 weeks.
  The participant tilted their head as far back as possible. Then, the researcher placed the goniometer's pivot point over the participant's ear, extending the goniometer over the tip of the participant's nose. Measure and record the data.

CONTACTS AND LOCATIONS:
Overall Officials: Wannaporn Tongtako, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No